CLINICAL TRIAL: NCT01444144
Title: Ankle Fracture Treatment in the Elderly, at Risk Population
Brief Title: Ankle Fracture Treatment in the Elderly
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 146-2011
Record Dates: First submitted 2011-09-26; First posted 2011-09-30 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Ankle Fracture
Keywords: Ankle; Fracture; Elderly; At-risk Population; Ankle Fracture in at-risk elderly population
MeSH Terms: conditions — Ankle Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankle Fracture: Patients aged 55 years at time of surgery undergoing treatment for ankle fractures.
  Interventions: Other: Fracture union

INTERVENTIONS:
Other: Fracture union — Retrospective records review post-operatively until fracture resolved.

SUMMARY:
The purpose of this study is to track surgical outcomes and post-operative course in patients 55 years of age or older treated for ankle fractures.

DETAILED DESCRIPTION:
This study seeks to describe and track surgical outcomes associated with the use of a minimally invasive surgical technique used to treat ankle fractures in at-risk patients 55 years of age or older

ELIGIBILITY:
Inclusion Criteria:

* at least 55 years of age at time of surgery
* receiving treatment for ankle fractures

Exclusion Criteria:

* none

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At-risk population, at least 55 years of age at time of surgery receiving treatment for ankle fractures.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-04-03 (Actual); Study Completion 2011-04-03 (Actual)

PRIMARY OUTCOMES:
Status of Fracture Union | Post-operatively until documentation of fracture healing, assessed up to seven months following surgery.
  Retrospective records review tracking ankle fractures post-operatively until fracture heals.

SECONDARY OUTCOMES:
Post-operative Complications | Post-operatively until documentation that complications resolved, assessed up to seven months following surgery.
  Retrospective record review tracking complications post-operatively until resolved.

CONTACTS AND LOCATIONS:
Overall Officials: Kalia K Sadasivan, M.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States